CLINICAL TRIAL: NCT03879655
Title: A Phase 2B/3 Open-label Trial of VTS-270 (2-hydroxypropyl-β-cyclodextrin) in Subjects With Neurologic Manifestations of Niemann-Pick Type C1 Disease Previously Treated Under Protocol VTS301
Brief Title: Open-label Study of VTS-270 in Participants With Neurologic Manifestations of Niemann-Pick Type C1
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated by previous Sponsor decision
Sponsor: Mandos LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTS-270-302
Record Dates: First submitted 2018-12-12; First posted 2019-03-19 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Niemann-Pick Disease, Type C
Keywords: Niemann-Pick; NPC
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — Cyclodextrins; 2-Hydroxypropyl-beta-cyclodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VTS-270 (Experimental): Eligible participants who transition into this study will receive treatment with VTS-270 at the last dose level administered in Study VTS301, administered IT via LP infusion every 2 weeks, for up to a total duration of 3 years or until the investigator considers VTS-270 to be no longer beneficial to the participant, VTS-270 receives marketing authorization, or the VTS-270 development program is discontinued.
  Interventions: Drug: VTS-270

INTERVENTIONS:
Drug: VTS-270 — Administered IT via LP infusion of VTS-270
  Other Names: 2-hydroxypropyl-β-cyclodextrin; Cyclodextrin; Adrabetadex

SUMMARY:
This is a multicenter, multinational, open-label study of VTS-270 to evaluate the long-term safety and tolerability of VTS-270 (2-hydroxypropyl-β-cyclodextrin) in participants transitioning from Study VTS301 (Parts A/B [NCT02534844] and Part C [NCT04958642]) with neurologic manifestations of Niemann-Pick Type C1 (NPC1) disease.

DETAILED DESCRIPTION:
Non-clinical studies and a Phase 1 clinical trial suggest that intrathecal (IT) administration of VTS-270 in participants with neurologic manifestations of NPC1 disease has the potential to slow the rate of progression of their neurologic disease. NPC1 disease is a rare, neurodegenerative, inherited, autosomal recessive lysosomal lipid storage disorder primarily in children and teenagers. The disease is characterized by the inability to properly metabolize cholesterol and other lipids within the cell due to mutations in the NPC1 gene causing unesterified cholesterol to accumulate in the brain, liver and spleen.

Eligible participants who transition into this study will receive treatment with VTS-270 at the last dose level administered in Study VTS301, administered IT via lumbar puncture (LP) infusion every 2 weeks, for up to a total duration of 3 years or until the investigator considers VTS-270 to be no longer beneficial to the participant, VTS-270 receives marketing authorization, or the VTS-270 development program is discontinued.

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible to participate in the study, at the Baseline Visit (except as noted below):

1. Participant completed Part B of Study VTS301 (defined as having completed Visit 27/Week 52 or completed at least through Visit 13/Week 24 and required rescue option) and is continuing in Part C of Study VTS301.
2. Participant, in the opinion of the Principal Investigator, should continue treatment with VTS-270.
3. Females of childbearing potential (not surgically sterile) must use a medically acceptable method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study. Acceptable methods of contraception include barrier method with spermicide, intrauterine device, steroidal contraceptive in conjunction with a barrier method, abstinence, or same-sex partner.
4. Participant or parent/guardian must provide written informed consent to participate in the study. In addition to parental consent, assent to participate must also be sought from minor children.

Key Exclusion Criteria:

A participant is ineligible for study participation if, at the Baseline Visit:

1. Participants discontinued from Study VTS301 for AEs.
2. Participant has an unresolved serious adverse event (SAE) for which treatment with VTS-270 has been halted.
3. Female participants who are pregnant or nursing.
4. Participants with suspected infection of the central nervous system or any systemic infection.
5. Participants with a spinal deformity that could impact the ability to perform a LP.
6. Participants with a skin infection in the lumbar region within 2 months of study entry.
7. Any of the following laboratory abnormalities at the Baseline Visit:

   1. Neutropenia, defined as an absolute neutrophil count of less than 1.5 × 10^9/liter (L).
   2. Thrombocytopenia (platelet count of less than 75 × 10^9/L).
   3. Activated partial thromboplastin time or prothrombin time prolonged by greater than 1.5 × the upper limit of normal (ULN) or known history of a bleeding disorder.
   4. Aspartate aminotransferase or alanine aminotransferase (ALT) greater than 4 × ULN.
   5. Anemia: hemoglobin greater than 2 standard deviations below normal for age and gender.
   6. Estimated glomerular filtration rate less than 60 milliliters (mL)/minute/1.73 square meter (m^2) calculated using the modified Schwartz formula (Schwartz et al., 2009) for participants aged 4 through 17 years old or using the Chronic Kidney Disease Epidemiology Collaboration equation formula for participants aged 18 years or older.
8. Evidence of obstructive hydrocephalus or normal pressure hydrocephalus.
9. Recent use of anticoagulants (in past 2 weeks prior to first dose [Study Day 0]).
10. Active pulmonary disease, oxygen requirement, or clinically significant history of decreased blood oxygen saturation, pulmonary therapy, or requiring active suction.
11. Participants who, in the opinion of the investigator, are unable to comply with the protocol or have medical conditions that would potentially increase the risk of participation.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Lead, Study Director — Mandos LLC
Locations (1):
- Hospital Clinica Biblica, San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included participants who completed Study VTS301 (Parts A/B [NCT02534844] and Part C [NCT04958642]) and were judged to receive potential benefit from continued treatment with adrabetadex. The study has been terminated early by the Sponsor due to previous Sponsor decision.
Groups:
- Adrabetadex: Participants received treatment with adrabetadex at the last dose level administered in Study VTS301, administered intrathecal (IT) via lumbar puncture (LP) infusion every 2 weeks, for up to a total duration of 3 years or until the investigator considered adrabetadex to be no longer beneficial to the participant, adrabetadex received marketing authorization, or the adrabetadex development program was discontinued.
Period: Overall Study
Arm/Group | Adrabetadex
Started | 2
Received at Least 1 Dose of Study Drug | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Adrabetadex: Participants received treatment with adrabetadex at the last dose level administered in Study VTS301, administered IT via LP infusion every 2 weeks, for up to a total duration of 3 years or until the investigator considered adrabetadex to be no longer beneficial to the participant, adrabetadex received marketing authorization, or the adrabetadex development program was discontinued.
Arm/Group | Adrabetadex
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No data is reported here to maintain participant confidentiality.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: No data is reported here to maintain participant confidentiality.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: No data is reported here to maintain participant confidentiality.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A TEAE was defined as an AE with onset on or after the start of adrabetadex treatment. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 156
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Adrabetadex
Number analyzed (Participants) | 2
Participants
  All TEAEs | 2
  SAEs | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 156
Description: All enrolled participants
Arm/Group | Adrabetadex
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adrabetadex (N=2)
Joint injury (Injury, poisoning and procedural complications) | 1
Influenza (Infections and infestations) | 1
Hypoacusis (Ear and labyrinth disorders) | 2
Asthenia (General disorders) | 1
Gelastic seizure (Nervous system disorders) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Dysphagia (Gastrointestinal disorders) | 1
Anal incontinence (Gastrointestinal disorders) | 1
Ataxia (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Hypokinesia (Nervous system disorders) | 1
Language disorder (Nervous system disorders) | 1
Anhedonia (Psychiatric disorders) | 1
Staring (Psychiatric disorders) | 1
Fatigue (General disorders) | 1
Seizure (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated by the Sponsor and only 2 participants were enrolled in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT03879655/Prot_SAP_001.pdf